CLINICAL TRIAL: NCT03200938
Title: Clinical Applicability of PBS® CIMMO Cement in Decoded Teeth Pulpotomies as Base and Restoration
Brief Title: Clinical Applicability of PBS® CIMMO Cement in Pulpotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, José Dias da Silva Neto, Clinical Professor, Principal Investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 57617816.9.0000.5102
Record Dates: First submitted 2017-05-03; First posted 2017-06-27 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Pulpotomy
Keywords: pulpotomy; Biological cement; Deciduous tooth

STUDY DESIGN:
Intervention Model Description: Comparative study with same series for the two groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blind study, the patient is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBS CIMMO (Experimental): Intervention: PBS CIMMO cement
  Interventions: Device: PBS CIMMO cement.
- Zinc oxide (Active Comparator): Intervention: Formocresol and zinc oxide
  Interventions: Device: formocresol and zinc oxide.

INTERVENTIONS:
Device: formocresol and zinc oxide. — Removal of the coronary pulp from primary molar teeth, use of formocresol and zinc oxide
  Other Names: Formocresol and zinc oxide technique
  Arms: Zinc oxide
Device: PBS CIMMO cement. — Removal of the coronary pulp from primary molar teeth, use of PBS cement
  Other Names: PBS CIMMO technique
  Arms: PBS CIMMO

SUMMARY:
Randomized clinical study in pulpotomies of deciduous molar teeth. A comparison of two techniques is established.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial conducted at the Universidade do Vale do Sapucaí (UNIVAS), Pouso Alegre, Minas Gerais and the University of Vale do Rio Verde (UNINCOR) Três Corações, Minas Gerais. A project will be submitted to the Brazil Platform to UNIVÁS and UNINCOR ethics committees. Thirty children aged four to ten years old will be selected from the Pediatric Dentistry Clinic of the College of Dentistry of the Vale do Rio Verde Três Corações University. The sample will consist of 30 primary molars that show indication for pulpotomy. The inclusion criteria of the teeth to be selected are: absence of spontaneous painful symptomatology in the preoperative period, evidence of live red bleeding, cut resistance, associated with hemostasis after exposure of the pulp tissue. Radiographically, the teeth should present 2/3 of the root length, absence of radiolucent inter-radicular lesion and internal root resorption.

The technique recommended will be in a single session. Local anesthesia with 1: 100,000 articaine (DFL®) will be used a tube containing 1.8 ml. Absolute insulation with clamp 14 (IVORY®), rubber sheet (Madeitex®) and arch (JON®). The opening will be performed with a 1016 HL (KG®) drill and a dentin curette (Duflex®). All carious tissue and the coronary pulp will be removed with abundant irrigation.

In group A (control) the irrigation will be with physiological saline and then it will be applied in the pulp chamber with autoclaved cotton ball, formocresol for five minutes. Subsequently, calcium hydroxide cement base (Hidro C®), zinc oxide cement base and eugenol (IRM®) and restoration of the final tooth with composite resin will be inserted.

In group B the irrigation will be with sterile distilled water (the cement to be used loses its properties in front of the saline solution). Excess blood and distilled water from the irrigation will be sucked through disposable endodontic cannula (DFL®) and the fast trapped PBS®CIMMO cement will be handled through sterile glass plate and spatula 24 (Duflex®). Then it will be taken to the humid chamber with cement door, old amalgam (Duflex®) and condenser with Schilder condenser number 5 (Odus®). The cement will serve as a sub-base, base and final restoration.

Patients will be submitted to final radiographs and receive systemic medication with analgesic and anti-inflammatory. The evaluations will be carried out in 6 months and will be through clinical and radiographic examinations, to define the result of the treatments. Clinical examinations will be performed under artificial light through an exploratory probe (Duflex®) and clinical mirror (Duflex®). The clinical criteria to be observed are: edema, mobility, fistula and pain. The radiographic evaluations will be through periapical radiography with the aid of a radial ortho positioner (DFL®). In the radiographs will be observed the presence or absence of internal and external resorptions, as well as presence or absence of inter-radicular lesion.

The statistical analysis will be through the chi-square test and the level of significance will be 5%.

ELIGIBILITY:
Inclusion criteria:

* Teeth exhibiting caries exposure
* Teeth with incomplete rhizogenesis
* Absence of periradicular lesion and fistula
* Accidental pulp exposure

Exclusion Criteria:

* Teeth with spontaneous pain
* Teeth With impossibility to perform absolute isolation
* Teeth with mobility, presence of fistula and root resorption of more than two-thirds of the root
* Teeth unable to be restored
* Teeth with painful response after vertical percussion

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Clinical examination evaluate the repair capacity of PBS® CIMMO and Zinc Oxide cements in pulpotomies will be evaluated. | 12 months
  The restorative capacity of the PBS CIMMO and Zinc Oxide cements will be assessed by clinical and radiographic examination six months after the pulpotomies.

SECONDARY OUTCOMES:
Radiografhic examination evaluate the repair capacity of PBS CIMMO and Zinc Oxide | 12 months
  The restorative capacity of CIMMO PBS and Zinc Oxide cements will be assessed by radiographic examination six months after pulpotomies.

CONTACTS AND LOCATIONS:
Overall Officials: José Neto, Principal Investigator — teacher
Locations (2):
- Brazil (2):
  - Fernanda Valadão Moysés, Pouso Alegre, Minas Gerais
  - Univás, Pouso Alegre, Minas Gerais

IPD SHARING:
Plan to Share IPD: No